CLINICAL TRIAL: NCT02289742
Title: Characterization of Pre-Lens Tear Film Stability of Daily Disposable Multifocal and Toric Contact Lenses Using Ring Mire Projection
Brief Title: Tear Film Evaluation of Dailies® AquaComfort Plus® Multifocal and Toric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: M-14-010
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Results first posted 2016-07-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-06

CONDITIONS: Refractive Error
Keywords: Dailies AquaComfort Plus® Multifocal (DACP MF); Dailies AquaComfort Plus® Toric (DACP Toric); tear film stability; Non-Invasive Keratograph Break-Up Time (NIK-BUT)
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm1: Presbyopes (Other): Nelfilcon A contact lenses (multifocal and sphere) worn as randomized in a crossover design during Periods 1 and 2, with nelfilcon A sphere contact lenses in Period 3. Each product worn bilaterally (in both eyes) for 12 hours.
  Interventions: Device: Nelfilcon A multifocal contact lenses; Device: Nelfilcon A sphere contact lenses
- Arm2: Astigmats (Other): Nelfilcon A contact lenses (toric and sphere) worn as randomized in a crossover design during Periods 1 and 2, with nelfilcon A sphere contact lenses in Period 3. Each product worn bilaterally (in both eyes) for 12 hours.
  Interventions: Device: Nelfilcon A toric contact lenses; Device: Nelfilcon A sphere contact lenses

INTERVENTIONS:
Device: Nelfilcon A multifocal contact lenses
  Other Names: DAILIES® AquaComfort Plus® Multifocal; DACP MF
  Arms: Arm1: Presbyopes
Device: Nelfilcon A toric contact lenses
  Other Names: DAILIES® AquaComfort Plus® Toric; DACP Toric
  Arms: Arm2: Astigmats
Device: Nelfilcon A sphere contact lenses
  Other Names: DAILIES® AquaComfort Plus®; DACP

SUMMARY:
The purpose of this study is to evaluate the pre lens tear film characteristics of DAILIES® Aqua Comfort Plus® Multifocal (DACP MF) and Toric (DACP Toric) compared to DAILIES® Aqua Comfort Plus® Sphere (DACP) daily disposable contact lenses over 12 hours of lens wear.

DETAILED DESCRIPTION:
Two population groups (presbyopes and astigmats) will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Must sign an informed consent document;
* Adapted, current soft contact lens wearer with either:

  1. A spectacle add between +0.50 and +2.50 (inclusive) [Presbyopes group]
  2. A spherical correction of an astigmatism up to 20% of the amount of the sphere [Astigmats group];
* Contact lens prescription in the power range specified in the protocol;
* Vision correctable to 0.2 logMAR (logarithmic minimal angle for resolution) or better in each eye at distance with pre-study lenses or manifest refraction at Visit 1;
* Willing to wear study lenses up to 12 hours and attend all study visits;
* Can be successfully fitted with study lenses;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Any ocular anterior segment infection, inflammation, abnormality, or active disease that would contraindicate contact lens wear;
* Use of systemic or ocular medications for which contact lens wear could be contraindicated as determined by the investigator;
* Use of artificial tears and rewetting drops during the study;
* Monocular (only 1 eye with functional vision) or fit with only 1 lens;
* Any abnormal ocular condition observed during the Visit 1 slit-lamp examination;
* History of herpetic keratitis, ocular surgery, or irregular cornea;
* Pregnant or lactating;
* Unstable tear film with a NIK-BUT value below 8 seconds in either eye without lenses;
* Participation in any clinical study within 30 days of Visit 1;
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Manager, Global Med Affairs, Operations, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 1 study center located in Germany.
Pre-assignment Details: Of the 48 enrolled subjects, 3 were discontinued as screen failures prior to randomization. This reporting group includes all randomized subjects (45).
Groups:
- Presbyopes MF/Sphere: Nelfilcon A multifocal contact lenses in Period 1, followed by nelfilcon A sphere contact lenses in Periods 2 and 3. Each product worn bilaterally (in both eyes) for 12 hours.
- Presbyopes Sphere/MF: Nelfilcon A sphere contact lenses in Periods 1 and 3, with nelfilcon A multifocal contact lenses in Period 2. Each product worn bilaterally (in both eyes) for 12 hours.
- Astigmats Toric/Sphere: Nelfilcon A toric contact lenses in Period 1, followed by nelfilcon A sphere contact lenses in Periods 2 and 3. Each product worn bilaterally (in both eyes) for 12 hours.
- Astigmats Sphere/Toric: Nelfilcon A sphere contact lenses in Periods 1 and 3, with nelfilcon A toric contact lenses in Period 2. Each product worn bilaterally (in both eyes) for 12 hours.
Period: First Wear Period
Arm/Group | Presbyopes MF/Sphere | Presbyopes Sphere/MF | Astigmats Toric/Sphere | Astigmats Sphere/Toric
Started | 11 | 12 | 12 | 10
Treated | 11 | 11 | 12 | 9
Completed | 11 | 11 | 11 | 9
Not Completed | 0 | 1 | 1 | 1
Not completed — Adverse event prior to treatment | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Other prior to treatment | 0 | 0 | 0 | 1
Period: Second Wear Period
Arm/Group | Presbyopes MF/Sphere | Presbyopes Sphere/MF | Astigmats Toric/Sphere | Astigmats Sphere/Toric
Started | 11 | 11 | 11 | 9
Completed | 11 | 11 | 11 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Third Wear Period
Arm/Group | Presbyopes MF/Sphere | Presbyopes Sphere/MF | Astigmats Toric/Sphere | Astigmats Sphere/Toric
Started | 11 | 11 | 11 | 9
Completed | 11 | 10 | 11 | 8
Not Completed | 0 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Reason not given | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized and exposed subjects.
Groups:
- Presbyopes: Nelfilcon A contact lenses (multifocal and sphere) worn as randomized in a crossover design during Periods 1 and 2, with nelfilcon A sphere contact lenses in Period 3. Each product worn bilaterally (in both eyes) for 12 hours.
- Astigmats: Nelfilcon A contact lenses (toric and sphere) worn as randomized in a crossover design during Periods 1 and 2, with nelfilcon A sphere contact lenses in Period 3. Each product worn bilaterally (in both eyes) for 12 hours.
- Total: Total of all reporting groups
Arm/Group | Presbyopes | Astigmats | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (8.1) | 25.8 (4.5) | 39.0 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  Germany | 22 | 21 | 43

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Wettability Grade of 2 or 3 After 12 Hours of Wear
Description: A video was made to capture a visual demonstration of tear film characteristics in between blinks. The investigator graded contact lens surface wettability using a scale from 0 (fully wettable) to 3 (clearly visible distortions) at 5, 10, 15, 20 and 25 seconds post-blink by region (central, superior, nasal, inferior, and temporal). Three independent measurements (3 blinks) were carried out. An average was taken over the 3 measurements, 5 regions, and 5 time points. One eye contributed to the analysis.
Time Frame: Hour 12, each product
Population: This analysis population includes all randomized and exposed subjects with data at visit.
Measure: Number; unit: percentage of subjects
Groups:
- Presbyopes / Multifocal: Nelfilcon A multifocal contact lenses worn bilaterally (in both eyes) for 12 hours during Period 1 or 2
- Presbyopes / Sphere: Nelfilcon A spherical contact lenses worn balaterally (in both eyes) for 12 hours during Period 1 or Period 2 (in a crossover design) and in Period 3
- Astigmats / Toric: Nelfilcon A toric contact lenses worn bilaterally (in both eyes) for 12 hours during Period 1 or Period 2 (in a crossover design)
- Astigmats / Sphere: Nelfilcon A spherical contact lenses worn bilaterally (in both eyes) for 12 hours during Period 1 or Period 2 (in a crossover design) and in Period 3
Arm/Group | Presbyopes / Multifocal | Presbyopes / Sphere | Astigmats / Toric | Astigmats / Sphere
Number analyzed (Participants) | 22 | 22 | 21 | 20
percentage of subjects | 55.8 | 47.2 | 46.5 | 49.5

2. Secondary Outcome: Percentage of Subjects With Wettability Grade of 2 or 3 After 8 Hours of Wear
Description: as for outcome 1
Time Frame: Hour 8, each product
Population: This analysis population includes all randomized and exposed subjects with data at visit.
Measure: Number; unit: percentage of subjects
Groups:
- Astigmats / Toric: Nelfilcon A toric contact lenses worn bilaterally (in both eyes) for 12 hours during Period 1 or Period 2 ( in a crossover design)
Arm/Group | Presbyopes / Multifocal | Presbyopes / Sphere | Astigmats / Toric | Astigmats / Sphere
Number analyzed (Participants) | 22 | 22 | 21 | 20
percentage of subjects | 60.8 | 46.3 | 34.3 | 33.3

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of a subject's participation in the study (up to 24 days). Ocular adverse events are presented for both study eye and non-study eye combined. AEs were reported as pre-treatment and treatment-emergent.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users or other persons, whether or not related to the medical device.
Groups:
- Pre-treatment: All subjects who consented to participate in the study prior to the initiation of study treatment
- Presbyopes / Multifocal: All subjects exposed to nelfilcon A multifocal contact lenses, worn bilaterally (in both eyes) for 12 hours during Periods 1 or 2 as randomized
- Presbyopes / Sphere First Exposure: All presbyopes exposed to nelfilcon A spherical contact lenses, worn bilaterally (in both eyes) for 12 hours during Period 1 or Period 2 as randomized
- Presbyopes / Sphere Second Exposure: All presbyopes exposed to nelfilcon A spherical contact lenses, worn bilaterally (in both eyes) for 12 hours during Period 3
- Astigmats / Toric: All subjects exposed to nelfilcon A toric contact lenses, worn bilaterally (in both eyes) for 12 hours during Periods 1 or 2 as randomized
- Astigmats / Sphere First Exposure: All astigmats exposed to nelfilcon A spherical contact lenses, worn bilaterally (in both eyes) for 12 hours during Period 1 or Period 2 as randomized
- Astigmats / Sphere Second Exposure: All astigmats exposed to nelfilcon A spherical contact lenses, worn bilaterally (in both eyes) for 12 hours during Period 3
Arm/Group | Pre-treatment | Presbyopes / Multifocal | Presbyopes / Sphere First Exposure | Presbyopes / Sphere Second Exposure | Astigmats / Toric | Astigmats / Sphere First Exposure | Astigmats / Sphere Second Exposure
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/22 | 0/22 | 0/22 | 0/21 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/48 | 0/22 | 0/22 | 0/22 | 0/21 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.